CLINICAL TRIAL: NCT01323270
Title: A Phase 2, Randomized, Placebo-controlled, Single-blind Trial To Assess The Safety, Tolerability, And Immunogenicity Of Repevax(Registered) And Bivalent Rlp2086 Vaccine When Administered Concomitantly In Healthy Subjects Aged Greater Than Or Equal To 11 To <19 Years
Brief Title: A Trial to Assess the Safety, Tolerability and Immunogenicity of Repevax and rLP2086 Vaccine When Given Together in Healthy Subjects Aged >=11 to <19 Years.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B1971010; 6108A1-2008 (Other: Alias Study Number); 2010-022449-38 (EudraCT Number)
Record Dates: First submitted 2011-02-17; First posted 2011-03-25 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Meningococcal Vaccine; rLP2086; Repevax; N Meningitidis Serogroup B; Meningitis
Keywords: Healthy adolescents
MeSH Terms: conditions — Meningitis | interventions — factor H-binding protein, Neisseria meningitidis; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rLP2086 (Experimental): rLP2086 and Repevax
  Interventions: Biological: rLP2086; Biological: Repevax
- Saline and Repevax (Placebo Comparator): Saline and Repevax
  Interventions: Biological: Saline; Biological: Repevax

INTERVENTIONS:
Biological: rLP2086 — 0.5 mL dose, given at 0, 2 and 6 months.
  Arms: rLP2086
Biological: Repevax — 0.5 mL dose, given at 0 months.
  Arms: rLP2086
Biological: Saline — 0.5 mL dose, given at 0, 2 and 6 months.
  Arms: Saline and Repevax
Biological: Repevax — 0.5 mL dose, given at 0 months.
  Arms: Saline and Repevax

SUMMARY:
This study is to look at a new vaccine that might prevent meningococcal disease, and to look at the safety of the new vaccine as well as how it is tolerated when given together with Repevax. The study will be done in healthy adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the parent/legally acceptable representative and/or subject has been informed of all pertinent aspects of the study.
* Parent/legally acceptable representative and/or subjects who are willing and able to comply with scheduled visits, laboratory tests, and other study procedures.
* Male or female subject aged ≥11 and <19 years at the time of enrollment.
* Available for the entire study period and can be reached by telephone.
* Healthy subject as determined by medical history, physical examination, and judgment of the investigator.
* Has received full series of diphtheria, tetanus, and pertussis (DTP)/DTaP vaccines and oral poliomyelitis virus (OPV)/IPV vaccines per country-specific recommendations applicable at the time of receipt.
* All male and female subjects must agree to practice a form of effective contraception, such as barrier contraception (ie, condom plus spermicide, a female condom, diaphragm, cervical cap or intrauterine device), implants, injectables, combined oral contraceptives or sexual abstinence prior to entering into the study, for the duration of the vaccination period and for 28 days after the last study vaccination. For Germany: The phrase sexual abstinence is not applicable, with the understanding that all male and all female subjects of childbearing potential must practice an effective form of contraception during the study.
* Negative urine pregnancy test for female subjects.

Exclusion Criteria:

* Previous vaccination with any meningococcal serogroup B vaccine.
* Vaccination with any diphtheria, tetanus, pertussis, or poliomyelitis virus vaccine within 5 years of the first study vaccination.
* A previous anaphylactic reaction to any vaccine or vaccine-related component.
* Contraindication to vaccination with diphtheria, tetanus, pertussis, or poliomyelitis virus vaccine.
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
* A known or suspected disease of the immune system or those receiving immunosuppressive therapy.
* History of culture-proven disease caused by Neisseria meningitidis or Neisseria gonorrhoeae.
* Significant neurological disorder or history of seizure (excluding simple febrile seizure).
* Receipt of any blood products, including immunoglobulin within 6 months before the first study vaccination.
* Current chronic use of systemic antibiotics.
* Participation in other studies during study participation. Participation in purely observational studies is acceptable.
* Received any investigational drugs, vaccines or devices within 28 days before administration of the first study vaccination.
* Any neuroinflammatory or autoimmune condition, including, but not limited to, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Subjects who are investigational site staff members or subjects who are Pfizer employees directly involved in the conduct of the trial.
* Subject is a direct descendant (eg, child, grandchild or other family member) of study site or Pfizer personnel.
* Subject is pregnant or breastfeeding.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 753 (Actual)
Dates: Start 2011-03-18 (Actual); Primary Completion 2012-10-08 (Actual); Study Completion 2013-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- Finland (14):
  - Espoo Vaccine Research Clinic, Espoo
  - Helsinki South Vaccine Research Clinic, Helsinki
  - Ita-Helsinki Vaccine Research Clinic, Helsinki
  - Järvenpää Vaccine Research Clinic, Jarvenpaa
  - Kokkola Vaccine Research Clinic, Kokkola
  - Lahti Vaccine Research Clinic, Lahti
  - Oulu Vaccine Research Clinic, Oulu
  - Pori Vaccine Research Clinic, Pori
  - Seinäjoki Vaccine Research Clinic, Seinäjoki
  - Tampereen Yliopisto University Of Tampere, Tampere
  - Tampere Vaccine Research Clinic, Tampere
  - Vaccine Research Center, Tampere
  - Turku Vaccine Research Clinic, Turku
  - Vantaa Vaccine Research Clinic, Vantaa
- Germany (10):
  - Gemeinschaftspraxis Dr. med. Guido Hein, Dr. med. Rainer Lauf, Bad Sobernheim
  - Gerhard Bleckmann Kinder- und Jugendarzt, Baunatal
  - Kinderarzt-Praxis, Bramsche
  - Gemeinschaftspraxis fuer Kinder- und Jugendmedizin Dres. Behre, Burgert, Gunkel, Kehl
  - Dr. med. Sobhi Mahdi Kinderarzt und Jugendmedizin, Lübeck
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Dr. Michael Vomstein, Hermann Oesterle, Kinder- und Jugendaerzte, Schwäbisch Hall
  - Thomas Lenz & (Frau) Dr. med. Marin Eggers, Vellmar
  - Dres.T. Schmitz, H. Knee, Ch, Wittermann Fachaerztliche, Weilheim
  - Gemeinschaftspraxis fuer Kinder und Jugendliche Welzheim, Welzheim
- Poland (12):
  - Gabinet Lekarski, Dębica
  - Krakowski Szpital Specjalistyczny, im. Jana Pawla II, Krakow
  - Specjalistyczna Praktyka Lekarska Gravita, Lodz
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Oddzial Pediatryczny, Lubartów
  - NZOZ Praktyka Lekarza Rodzinnego Eskulap, Lublin
  - NZOZ Praktyka Lekarza Rodzinnego Alina Grocka-Wlazlak, Oborniki Śląskie
  - Specjalistyczny ZOZ nad Matka i Dzieckiem, Przychodnia Wieku Rozwojowego, Poznan
  - NZLA Michalkowice Jarosz i Partnerzy, Siemianowice Śląskie
  - NZOZ Nasz Lekarz, Torun
  - Szpital im. Sw. Jadwigi Slaskiej, Oddzial Pediatryczny, Trzebnica
  - Samodzielny Publiczny Szpital Kliniczny nr 1 we Wroclawiu, Wroclaw
  - NZOZ Salmed, Łęczna

REFERENCES:
- [Derived] Beeslaar J, Mather S, Absalon J, Eiden JJ, York LJ, Crowther G, Maansson R, Maguire JD, Peyrani P, Perez JL. Safety data from the MenB-FHbp clinical development program in healthy individuals aged 10 years and older. Vaccine. 2022 Mar 15;40(12):1872-1878. doi: 10.1016/j.vaccine.2022.01.046. Epub 2022 Feb 11. PMID 35164991
- [Derived] Beeslaar J, Peyrani P, Absalon J, Maguire J, Eiden J, Balmer P, Maansson R, Perez JL. Sex, Age, and Race Effects on Immunogenicity of MenB-FHbp, A Bivalent Meningococcal B Vaccine: Pooled Evaluation of Clinical Trial Data. Infect Dis Ther. 2020 Sep;9(3):625-639. doi: 10.1007/s40121-020-00322-5. Epub 2020 Jul 17. PMID 32681472
- [Derived] Vesikari T, Wysocki J, Beeslaar J, Eiden J, Jiang Q, Jansen KU, Jones TR, Harris SL, O'Neill RE, York LJ, Perez JL. Immunogenicity, Safety, and Tolerability of Bivalent rLP2086 Meningococcal Group B Vaccine Administered Concomitantly With Diphtheria, Tetanus, and Acellular Pertussis and Inactivated Poliomyelitis Vaccines to Healthy Adolescents. J Pediatric Infect Dis Soc. 2016 Jun;5(2):180-7. doi: 10.1093/jpids/piv064. Epub 2016 Jan 23. PMID 26803328

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 753 participants were enrolled in this study. Of these, 4 participants were not randomized but were vaccinated rLP2086 vaccine or Repevax or Saline at Vaccination 1. These participants were included in safety population and not intent-to-treat population.
Groups:
- Group 1: rLP2086 + Repevax: Randomized to receive rLP2086 at 0-,2-6-month and Repevax at 0-month.
- Group 2: Saline+Repevax: Randomized to receive Saline at 0-,2-6-month and Repevax at 0-month.
Period: Overall Study
Arm/Group | Group 1: rLP2086 + Repevax | Group 2: Saline+Repevax
Started | 373 | 376
Completed | 330 | 347
Not Completed | 43 | 29
Not completed — Withdrawal by Subject | 19 | 10
Not completed — Protocol Violation | 9 | 7
Not completed — Lost to Follow-up | 4 | 6
Not completed — Adverse Event | 8 | 0
Not completed — Other | 0 | 3
Not completed — Physician Decision | 0 | 2
Not completed — Not eligible | 1 | 1
Not completed — Death | 1 | 0
Not completed — Randomized, but not vaccinated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: rLP2086 + Repevax | Group 2: Saline+Repevax | Total
Number analyzed (Participants) | 373 | 376 | 749
Age, Customized [Number; unit: participants]
  Greater than or equal (>=)11-less than (<)14years | 217 | 215 | 432
  >=14 years-<19 years | 156 | 161 | 317
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 184 | 367
  Male | 190 | 192 | 382

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Prespecified Criteria for the Concomitant Antigen
Time Frame: 1 month after Vaccination 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: rLP2086 + Repevax | Group 2: Saline+Repevax
Number analyzed (Participants) | 337 | 348
percentage of participants
  Diphtheria | 99.4 | 99.4
  Tetanus | 100.0 | 100.0
  Pertussis toxoid | 94.7 | 96.0
  Pertussis filamentous hemagglutinin | 100.0 | 100.0
  Pertussis pertactin | 100.0 | 100.0
  Pertussis fimbrial agglutinogens types 2+3 | 97.6 | 98.9
  Poliovirus type 1 | 100.0 | 100.0
  Poliovirus type 2 | 100.0 | 100.0
  Poliovirus type 3 | 100.0 | 100.0
Statistical Analysis 1: Comparison: Group 1: rLP2086 + Repevax vs Group 2: Saline+Repevax; Diphtheria: Exact 2-sided confidence interval (based on Chan and Zhang) was reported for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 10%; Percent difference = -0.0, 95% CI 2-sided [-1.6 to 1.5]
Statistical Analysis 2: Comparison: Group 1: rLP2086 + Repevax vs Group 2: Saline+Repevax; Tetanus: Exact 2-sided confidence interval (based on Chan and Zhang) was reported for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 10%; Percent difference = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 3: Comparison: Group 1: rLP2086 + Repevax vs Group 2: Saline+Repevax; Pertussis toxoid: Exact 2-sided confidence interval (based on Chan and Zhang) was reported for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 10%; Percent difference = -1.3, 95% CI 2-sided [-4.7 to 1.9]
Statistical Analysis 4: Comparison: Group 1: rLP2086 + Repevax vs Group 2: Saline+Repevax; Pertussis filamentous hemagglutinin: Exact 2-sided confidence interval (based on Chan and Zhang) was reported for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 10%; Percent difference = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 5: Comparison: Group 1: rLP2086 + Repevax vs Group 2: Saline+Repevax; Pertussis pertactin: Exact 2-sided confidence interval (based on Chan and Zhang) was reported for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 10%; Percent difference = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 6: Comparison: Group 1: rLP2086 + Repevax vs Group 2: Saline+Repevax; Pertussis fimbrial agglutinogens types 2+3: Exact 2-sided confidence interval (based on Chan and Zhang) was reported for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 10%; Percent difference = -1.2, 95% CI 2-sided [-3.6 to 0.8]
Statistical Analysis 7: Comparison: Group 1: rLP2086 + Repevax vs Group 2: Saline+Repevax; Poliovirus type 1: Exact 2-sided confidence interval (based on Chan and Zhang) was reported for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 10%; Percent difference = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 8: Comparison: Group 1: rLP2086 + Repevax vs Group 2: Saline+Repevax; Poliovirus type 2: Exact 2-sided confidence interval (based on Chan and Zhang) was reported for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 10%; Percent difference = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 9: Comparison: Group 1: rLP2086 + Repevax vs Group 2: Saline+Repevax; Poliovirus type 3: Exact 2-sided confidence interval (based on Chan and Zhang) was reported for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 10%; Percent difference = 0.0, 95% CI 2-sided [-1.1 to 1.1]

2. Secondary Outcome: Geometric Mean Concentration (GMC) for Diphtheria and Tetanus Antigens
Time Frame: 1 month after Vaccination 1
Measure: Geometric Mean (95% Confidence Interval); unit: International Units per milliliter
Arm/Group | Group 1: rLP2086 + Repevax | Group 2: Saline+Repevax
Number analyzed (Participants) | 337 | 348
International Units per milliliter
  Diphtheria | 1.4 [1.28 to 1.55] | 1.5 [1.34 to 1.63]
  Tetanus | 12.3 [11.50 to 13.11] | 12.4 [11.52 to 13.25]

3. Secondary Outcome: GMC for Acellular Pertussis Antigens
Description: Enzyme-linked immunosorbent assay (ELISA) units per milliliter (EU/mL)
Time Frame: 1 month after Vaccination 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: rLP2086 + Repevax | Group 2: Saline+Repevax
Number analyzed (Participants) | 337 | 348
EU/mL
  Pertussis toxoid | 27.1 [24.45 to 30.07] | 26.5 [23.95 to 29.38]
  Pertussis filamentous hemagglutinin | 119.4 [111.15 to 128.17] | 122.9 [115.14 to 131.13]
  Pertussis pertactin | 317.0 [285.64 to 351.80] | 336.1 [305.82 to 369.30]
  Pertussis fimbrial agglutinogens types 2+3 | 339.1 [296.35 to 387.94] | 364.5 [320.62 to 414.42]

4. Secondary Outcome: Geometric Mean Titer (GMT) for Poliomyelitis Antigens
Time Frame: 1 month after Vaccination 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: rLP2086 + Repevax | Group 2: Saline+Repevax
Number analyzed (Participants) | 337 | 348
titer
  Poliovirus type 1 | 662.1 [567.36 to 772.67] | 672.6 [581.87 to 777.55]
  Poliovirus type 2 | 840.5 [725.11 to 974.29] | 995.8 [860.54 to 1152.41]
  Poliovirus type 3 | 2237.4 [1945.81 to 2572.65] | 2450.1 [2152.60 to 2788.70]

5. Secondary Outcome: Percentage of Participants Achieving Serum Bactericidal Assay Using Human Complement (hSBA) Titer Level Greater Than or Equal to (>=) Prespecified Titer Level
Time Frame: 1 month after Vaccination 3
Population: Serum samples from approximately 50% of the participants had hSBA performed with primary MnB test strains expressing rLP2086 variants A22 and B24 and the other 50% of participants had hSBAs performed with strains expressing variants A56 and B44. The number of participants shown for each test strain represents the number with valid and determinant assay result for that strain.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: rLP2086 + Repevax | Group 2: Saline+Repevax
Number analyzed (Participants) | 307 | 330
percentage of participants
  PMB80 [A22] 1:16 (N=158, 166): number analyzed (Participants) | 158 | 166
  PMB80 [A22] 1:16 (N=158, 166) | 95.6 | 19.9
  PMB2001 [A56] 1:8 (N=148, 152): number analyzed (Participants) | 148 | 152
  PMB2001 [A56] 1:8 (N=148, 152) | 100.0 | 26.3
  PMB2948 [B24] 1:8 (N=157, 170): number analyzed (Participants) | 157 | 170
  PMB2948 [B24] 1:8 (N=157, 170) | 96.8 | 12.9
  PMB2707 [B44] 1:8 (N=146, 159): number analyzed (Participants) | 146 | 159
  PMB2707 [B44] 1:8 (N=146, 159) | 81.5 | 8.2

6. Other Pre Specified Outcome: Immunoglobulin G (IgG) Measured by Geometric Mean Titer (GMT)
Time Frame: Before vaccination 1, 1 month after Vaccination 2, 3
Population: A decision was made, a priori, that the hSBA MnB immunogenicity assay will be used instead of the IgG assay originally planned . Therefore only hSBA assay results will be disclosed.
Arm/Group | Group 1: rLP2086 + Repevax | Group 2: Saline+Repevax
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Geometric Mean Fold-Rise (GMFR) for IgG
Time Frame: Before Vaccination 1, 1 month after Vaccination 2, 3
Population: as for outcome 6
Arm/Group | Group 1: rLP2086 + Repevax | Group 2: Saline+Repevax
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Percentage of Participants With at Least One Adverse Event (AE)
Time Frame: Vaccination 1 up to 1 month after Vaccination 3
Population: Summary was performed for participants as per vaccine administration.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: rLP2086 + Repevax | Group 2: Saline+Repevax
Number analyzed (Participants) | 374 | 378
percentage of participants | 37.4 | 40.2

ADVERSE EVENTS:
Time Frame: AE reported from Vaccination 1 to 1 month after last administration of investigational product (bivalent rLP2086/saline/Repevax). SAE reported from Vaccination 1 to 6 months after last of investigational product (bivalent rLP2086/saline/Repevax).
Description: Events collected on case report form were reported. Summary was performed for participants as per vaccine administration.
Arm/Group | Group 1: rLP2086 + Repevax | Group 2: Saline+Repevax
Serious Adverse Events (participants affected / at risk) | 12/374 | 9/378
Other Adverse Events (participants affected / at risk) | 98/374 | 118/378
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: rLP2086 + Repevax (N=374) | Group 2: Saline+Repevax (N=378)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Syndactyly (Congenital, familial and genetic disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2
Abdominal abscess (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Drug abuse (Psychiatric disorders) | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: rLP2086 + Repevax (N=374) | Group 2: Saline+Repevax (N=378)
Conjunctivitis (Eye disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 1 | 4
Pyrexia (General disorders) | 5 | 4
Injection site pain (General disorders) | 4 | 0
Injection site swelling (General disorders) | 4 | 0
Nasopharyngitis (Infections and infestations) | 30 | 31
Pharyngitis (Infections and infestations) | 17 | 19
Upper respiratory tract infection (Infections and infestations) | 16 | 19
Bronchitis (Infections and infestations) | 9 | 18
Gastroenteritis (Infections and infestations) | 8 | 11
Sinusitis (Infections and infestations) | 8 | 6
Otitis media (Infections and infestations) | 3 | 7
Acute tonsillitis (Infections and infestations) | 1 | 7
Tonsillitis (Infections and infestations) | 1 | 7
Rhinitis (Infections and infestations) | 2 | 4
Contusion (Injury, poisoning and procedural complications) | 4 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 7
Headache (Nervous system disorders) | 9 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.